CLINICAL TRIAL: NCT04391218
Title: Applicabilità ed Efficacia di un Approccio Multi-Disciplinare Comprendente un Sistema Informatico di Supporto Per la Decisione Della Terapia di Pazienti Anziani Polipatologici
Brief Title: A Multidisciplinary Intervention Including a Clinical Decision Support System and an App for Drug Therapy Management in Older Patients
Acronym: FARMA-CANP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: University of Turin, Italy (Other); Infologic S.r.l., Padova, Italy (Unknown); Consoft Sistemi S.p.A. Turin, Italy (Unknown); ASL Città di Torino, Italy (Unknown)
Responsible Party: Principal Investigator, Dott.ssa RENATA MARINELLO, Dirigente Medico, S.C. Geriatria e Malattie Metaboliche dell'Osso U, Ospedalizzazione a Domicilio, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FARMA-CANP
Record Dates: First submitted 2020-05-06; First posted 2020-05-18 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Polypharmacy; Multimorbidity; Aged
Keywords: Clinical Decision Support System; App; Medication Adherence; Medication Reconciliation; Pharmacist; Inappropriate prescribing
MeSH Terms: conditions — Alzheimer Disease; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary Approach Group (Experimental): Multidisciplinary medication review and reconciliation during hospitalization involving geriatricians, nurses, pharmacists and supported by a Clinical Decision Support System, followed by an end-user App to support patients/caregivers in the correct drug intake after discharge.
  Interventions: Other: Multidisciplinary Approach Group
- Control Group (No Intervention): Medication review and reconciliation will be performed by geriatricians according to Good Clinical Practice and usual habits, that might also include digital and printed supports for medication appropriateness and drug interaction. Drug therapy will be listed and explained to the patient/caregiver at discharge. Patients/caregivers will be allowed to use any tools to support medication adherence, according to their habits and preferences (i.e. calendars, alarms, pill boxes).

INTERVENTIONS:
Other: Multidisciplinary Approach Group — Geriatricians will introduce medication review data on a Clinical Decision Support System, that will help both pharmacists and physicians in medication reconciliation, highligting potentially inappropriate prescriptions according to Beers' criteria and STOPP/START criteria, and potential controindicated and major Drug-Drug Interactions according to Micromedex. Before Hospital at Home discharge, nurses will instruct patients and/or caregivers to the use of an App, where daily drug therapy at discharge will be inserted and scheduled. This App will automatically create an alert everytime a drug dose needs to be taken, alongside an image of the specific drug packaging. The App will register if and when the patient actually takes the drug, or the reason for the delayed/missed dose.
  Arms: Multidisciplinary Approach Group

SUMMARY:
"La Casa nel Parco" (CANP) Project is a European Union and Regione Piemonte funded multidisciplinary project aimed to explore innovative technology application in older subject care. In this context, FARMA-CANP is a randomized open-label clinical trial evaluating a multidisciplinary intervention in older patients hospitalized at home. The intervention involves physicians, pharmacists, nurses and includes a Clinical Decision Support System to help the processes of therapeutic review and reconciliation, and an end-user App to support patients and/or caregivers in the daily management of drug therapy.

The main objectives of the study are to evaluate the impact of the intervention on 1) medication adherence after discharge 2) medication appropriateness.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 65 years
* Hospital at Home admission
* Presence of a caregiver
* Written informed consent signed by both the patient and the caregiver

Exclusion Criteria:

* Unavailable internet access and/or portable device to install the App on
* Severe cognitive impairment with behavioural symptoms
* Estimated life expectancy less than 3 months
* Death during Hospital at Home stay
* Hospital at Home discharge to an other healthcare facility (i.e. Emergency Department, Nursing Home)
* No regular medications precribed at Hospital at Home discharge.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a therapeutic adherence index ≥0.8 | 6 months after Hospital at Home discharge
  The therapeutic adherence index is defined as the ratio of number of drug units dispensed on total number of drug units prescribed at discharge.
  Data on drug units dispensed will be derived from a central database of territorial pharmaceutical center of A.S.L.Città di Torino.

SECONDARY OUTCOMES:
Number of Potentially Inappropriate Prescriptions (PIP) and number of participants with at least one Beers' PIP | At Hospital at Home discharge, an average of 14 days after group allocation
  Beers' PIPs will be identified according to the Beers' 2019 Criteria
Number of Potentially Inappropriate Prescriptions (PIP) and number of participants with at least one Screening Tool of Older People's Prescriptions (STOPP) PIP | At Hospital at Home discharge, an average of 14 days after group allocation
  STOPP IPs will be identified according to the Screening Tool of Older People's Prescriptions version 2
Number of potential contraindicated and/or major Drug-Drug Interactions (DDI) and number of participants with at least one potential contraindicated and/or major DDI. | At Hospital at Home discharge, an average of 14 days after group allocation
  Potential contraindicated and major DDIs will be identified using the Micromedex database

CONTACTS AND LOCATIONS:
Overall Officials: Renata Marinello, MD, PhD, Principal Investigator — A.O.U. Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] By the 2019 American Geriatrics Society Beers Criteria(R) Update Expert Panel. American Geriatrics Society 2019 Updated AGS Beers Criteria(R) for Potentially Inappropriate Medication Use in Older Adults. J Am Geriatr Soc. 2019 Apr;67(4):674-694. doi: 10.1111/jgs.15767. Epub 2019 Jan 29. PMID 30693946
- See also: Micromedex® online database. International Business Machines Corporation (IBM) Watson Health, Greenwood Village, Colorado, USA. — https://www.micromedexsolutions.com